CLINICAL TRIAL: NCT01928667
Title: Risk Factors for Microscopic Colitis: A Dutch Case-Control Study
Brief Title: Case-Control Study to Identify Risk Factors for Microscopic Colitis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL44127.068.13
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Microscopic Colitis; Collagenous Colitis; Lymphocytic Colitis
MeSH Terms: conditions — Colitis, Microscopic; Colitis, Collagenous; Colitis, Lymphocytic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — saliva samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Microscopic Colitis: Group consists of subjects diagnosed with either collagenous of lymphocytic colitis between January 1, 2000 and December 31, 2012
  Interventions: Other: Whole saliva sample
- Healthy Controls: Control group consists of subjects with no history of microscopic colitis. Group is age and sex matched with the case-group
  Interventions: Other: Whole saliva sample

INTERVENTIONS:
Other: Whole saliva sample — Both case and control group will be approached to consider to give permission to sample saliva. This is not obligatory. Collected samples will be stored for future DNA research.

SUMMARY:
The purpose of the study is to assess among others environmental and hygiene-related risk factors for microscopic colitis (MC), a common diarrheal disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of MC (CC or LC) between January 1, 2000 and December 31, 2012.
* Inhabitant of the province of Limburg or the Eindhoven region at the moment of diagnosis

Exclusion Criteria:

* Below 18 years of age at the time of diagnosis
* Not capable of signing an informed consent
* Deceased at moment of approximation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The case group will be selected by a retropective search in the pathology registry. Subjects have to be diagnosed between January 1, 2000 and December 31, 2012; have to be older than 18 years of age and have to be living in the province of Limburg, the Netherlands.
  Healthy controls are selected via the municipal personal records databases in the same region.
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Assessment of environmental and hygiene-related risk factors for microscopic colitis | Retrospective, between 2000 and 2012
  Information about environmental and hygiene-related risk factors is obtained by a questionnaire, sent to subjects diagnosed with MC between 2000 and 2012

SECONDARY OUTCOMES:
The difference between the CC and LC subpopulation regarding environmental, hygiene-related, and generally known risk factors | Retrospective between 2000 and 2012
  As generally known risk factors are considered: age, gender, medication, comorbidities and smoking.
  Information about risk factors is obtained by a questionnaire, sent to subjects diagnosed with MC between 2000 and 2012.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke J Pierik, MD, PhD, Principal Investigator — Maastricht UMC; Daisy MAE Jonkers, PhD, Principal Investigator — Maastricht University; Ad AM Masclee, Prof., Study Director — Maastricht UMC
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands